CLINICAL TRIAL: NCT06151821
Title: Examining the Influence of Guided Meditation on Diabetes-related Distress and Glycemic Control: A Randomized Controlled Trial Among Hospitalized Type 1 Adolescent Diabetic Patients
Brief Title: Examining the Influence of Guided Meditation on Diabetes-related Distress and Glycemic Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shifa International Hospital (Other)
Responsible Party: Principal Investigator, Saima Abass Tahammal, Principal Investigator, Shifa International Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SH-34988383
Record Dates: First submitted 2023-08-02; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 diabetes mellitus; Guided meditation; Adolescents
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor did not know which patients received the intervention and which patients did not
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group MTG (Experimental): The intervention arm received Guided Meditation sessions
  Interventions: Behavioral: Guided meditation
- Group STG (No Intervention): The control arm received standard care without any Guided meditation sessions

INTERVENTIONS:
Behavioral: Guided meditation — Meditation with guidance
  Arms: Group MTG

SUMMARY:
The study aims to investigate the effects of Guided Meditation on diabetes-related distress and glycemic control in hospitalized Type 1 adolescent diabetic patients. The study will employ a randomized controlled trial design, with participants randomly assigned to either the intervention group (receiving Guided Meditation sessions) or the control group (receiving standard care). The primary outcomes measured will be diabetes-related distress levels and glycemic control (HbA1c levels).

DETAILED DESCRIPTION:
The researchers hypothesize that the intervention group will experience a reduction in diabetes-related distress and an improvement in glycemic control compared to the control group. The study's findings could suggest how guided meditation could help manage the emotional distress and enhance diabetes management in hospitalized Type 1 adolescent diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent patients aged between 12 to 18 years.
* Confirmed diagnosis of Type 1 diabetes mellitus.
* Hospitalized in the participating medical facility.
* Capable of providing informed consent (for participants aged 18) or providing assent with parental/legal guardian consent (for participants aged 12 to 17).

Exclusion Criteria:

* Presence of severe psychiatric disorders or cognitive impairments that may hinder participation in the guided meditation sessions.
* Physical limitations or medical conditions that prevent the safe participation in the intervention or assessment procedures.
* Previously engaged in regular meditation or mindfulness practices, which may confound the results.
* Inability to communicate effectively in the language used for assessments and interventions.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-03 (Actual)

PRIMARY OUTCOMES:
Diabetes distress scale | Week 1 and Week 13
  Diabetes distress scale questionnaire

SECONDARY OUTCOMES:
HbA1c levels | Week 1 and Week 13
  HbA1c levels
Number of hypoglycemic and hyperglycemic episodes | Week 1, 4, 8 and 12
  Number of hypoglycemic and hyperglycemic episodes

CONTACTS AND LOCATIONS:
Overall Officials: Saima Abbass, MD, MSc, Principal Investigator — Shifa hospital
Locations (1):
- Shifa Hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No